CLINICAL TRIAL: NCT03003273
Title: Early Stoppage Versus Continuation of Antimicrobial Therapy in Low Risk Pediatric Cancer Patients With Febrile Neutropenia, Before Recovery of Counts: a Randomized Controlled Study -DALFEN Study
Brief Title: Early Stoppage Versus Continuation of Antimicrobial Therapy in Low Risk Pediatric Cancer Patients With Febrile Neutropenia, Before Recovery of Counts: -DALFEN Study
Acronym: DALFEN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, AKASH KUMAR, Senior Resident (DM course), All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IECPG-164
Record Dates: First submitted 2016-12-13; First posted 2016-12-28 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Neutropenia, Febrile; Pediatric Cancer
MeSH Terms: conditions — Febrile Neutropenia; Neoplasms | interventions — Amoxicillin-Potassium Clavulanate Combination; Levofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm (A) - stoppage of antibiotics (Experimental): patients will be reassessed for randomization once they fulfill all inclusion criteria and get afebrile for at least 24 hours. Antibiotics will be stopped in Arm-A.
  Interventions: Other: stoppage of antibiotics
- arm (B) - oral antibiotics till ANC ≥ 500 (Active Comparator): patients will be reassessed for randomization once they fulfill all inclusion criteria and get afebrile for at least 24 hours. oral antibiotics, in place of intravenous antibiotics, will be started in Arm-B.
  Interventions: Other: amoxycillin/clavulanic acid; Other: levofloxacin

INTERVENTIONS:
Other: stoppage of antibiotics — antibiotics will be stopped in arm - A on randomization, once child is afebrile for at least 24 hours and fulfills the inclusion criteria.
  Arms: arm (A) - stoppage of antibiotics
Other: amoxycillin/clavulanic acid — In arm - B, once the child is randomized, oral antibiotics will be started (Amoxicillin/ Clavulanic acid + Levofloxacin)
  Arms: arm (B) - oral antibiotics till ANC ≥ 500
Other: levofloxacin — In arm - B, once the child is randomized, oral antibiotics will be started (Amoxicillin/ Clavulanic acid + Levofloxacin)
  Arms: arm (B) - oral antibiotics till ANC ≥ 500

SUMMARY:
Pediatric patients with febrile neutropenia coming to Department of Medical Oncology with low risk features (culture awaited), will be started on intravenous antibiotics (Inj Cefoperazone+ Sulbactam ± Amikacin) on outpatient basis. Those patients will be reassessed for randomization once they fulfill all inclusion criteria and get afebrile for at least 24 hours. Antibiotics will be stopped in Arm-A and oral antibiotics, in place of intravenous antibiotics, will be started in Arm-B. The patients will be followed-up till ANC≥ 500, or reappearance of fever within follow-up of ≤ 10 days.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric febrile neutropenia patients treated on outpatient basis
* Age 3 years - 18 years
* Fulfilling low risk criteria ( Hematological malignancies in remission, No identifiable focus of infection, No Pneumonia/ mucositis / GI sepsis / Nausea-vomiting/ neurologic-mental status changes/ Central Venous Catheter (CVC) related infection, Anticipated Absolute Neutrophil Count (ANC) recovery ≤ 10 days, No organ dysfunction, Hemodynamically stable, Culture negative )
* Afebrile for at least 24 hours, on intra-venous antibiotics

Exclusion Criteria:

* Bone marrow involvement in solid tumor
* Already enrolled once, in previous episode
* On antibiotics prophylaxis
* Retroviral positive patients
* Patient undergone stem cell transplant

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Treatment is considered to be successful if the following is attained without changing the regimen - Patient remains afebrile till recovery of ANC ≥500 •Measure of effect: Proportion of patients afebrile in each arm | till ANC ≥ 500 or reappearance of fever during the period ≤ 10 days

SECONDARY OUTCOMES:
Rate of re-admission | till ANC ≥ 500 or reappearance of fever during the period ≤10 days

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Bakhshi, Professor, Study Director — Department of Medical Oncology, 2nd Floor, B.R.A.I.R.C.H, All India Institute of Medical Sciences, New Delhi, India
Locations (1):
- Department of Medical Oncology, AIIMS, New Delhi, India